CLINICAL TRIAL: NCT00412828
Title: A Phase I/II Study of CR011-vcMMAE in Subjects With Unresectable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CuraGen Corporation (Industry)
Responsible Party: Sponsor
Organization: Celldex Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011-CLN-11
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Unresectable Stage III or Stage IV Melanoma
Keywords: Melanoma; CR011-vcMMAE
MeSH Terms: conditions — Melanoma | interventions — CR011-vcMMAE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CR011-vcMMAE — administered as an intravenous infusion of 250 mL over 90 min

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of CR011-vcMMAE in patients who have unresectable stage III or stage IV melanoma and have failed no more than 1 line of prior cytotoxic therapy. CR011-vcMMAE will be administered intravenously (IV) once every 3 weeks at escalating doses until the maximum tolerated dose (MTD) is reached. Once the MTD is defined, 18-32 patients will be enrolled to further evaluate the safety and efficacy of CR011-vcMMAE at this dose level. Additional dosing schedules of CR011-vcMMAE will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age ≥ 18 years.
* Progressive or new metastatic melanoma, stage III or IV.
* Measurable disease by CT / MRI
* Failure of no more than 1 line of prior cytotoxic therapy.
* Adequate bone marrow, renal and hepatic function

  * Leukocytes ≥ 3000/mm3, ANC ≥ 1,500 cells/mm3, Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 10 g/dL (transfusion allowed)
  * Total bilirubin ≤ 1.5 x upper normal limit (UNL)
  * AST (SGOT), ALT (SGPT) ≤ 3.0 x UNL (≤ 5.0 x UNL may be acceptable)
  * Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance > 45 mL/min/1.73 m2
  * PT/aPTT < 1.5 x UNL or within therapeutic range via anti-coagulation therapy
* Karnofsky PS ≥ 70%.
* Estimated life expectancy > 3 months.
* Signed informed consent approved IRB and ability to comply with the study or monitoring procedures.
* Subjects with evaluable disease are eligible in dose-escalation cohorts

Exclusion Criteria:

* Prior therapies for disease under study less than 4 weeks prior to enrollment.
* Major surgery or trauma within 4 weeks of enrollment.
* Active brain metastases
* Active chronic inflammatory, autoimmunity, immunodeficiency disease, and vascular or hemorrhagic disorders.
* History of allergic reactions to dolastatin, auristatin or compounds of similar composition.
* Significant cardiovascular disease
* Other malignancies
* Pregnancy or breast feeding
* Refusal or inability to use effective means of contraception (for men, and women with childbearing potential)
* History of or test-positive to HIV, or hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
to evaluate the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) | throughout the study

SECONDARY OUTCOMES:
to evaluate the immune response to CR011-vcMMAE | throughout the study
to assess the pharmacodynamics and pharmacokinetics of CRO11-vcMMAE | throughout the study
to explore clinical anti-tumor response of CR011-vcMMAE in subjects with advanced metastatic melanoma | throughout the study

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Angeles Clinic and Research Institute, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - New York University Medical Center, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Ott PA, Hamid O, Pavlick AC, Kluger H, Kim KB, Boasberg PD, Simantov R, Crowley E, Green JA, Hawthorne T, Davis TA, Sznol M, Hwu P. Phase I/II study of the antibody-drug conjugate glembatumumab vedotin in patients with advanced melanoma. J Clin Oncol. 2014 Nov 10;32(32):3659-66. doi: 10.1200/JCO.2013.54.8115. Epub 2014 Sep 29. PMID 25267741
- See also: Phase I/II study of the antibody-drug conjugate glembatumumab vedotin in patients with advanced melanoma. — http://www.ncbi.nlm.nih.gov/pubmed/25267741